CLINICAL TRIAL: NCT00248703
Title: Secondary Adjuvant (Rescue) Treatment With Docetaxel (Taxotere) and Detection of Isolated Tumor Cells in Bone Marrow as a Surrogate Marker for Effect in Node Positive and High Risk Node Negative Breast Cancer After Standard Adjuvant Epirubicin-containing Treatment
Brief Title: Secondary Adjuvant Treatment for Patients With Isolated Tumor Cells in Bone Marrow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Tromso (Other); Helse Stavanger HF (Other Government); Sorlandet Hospital HF (Other Government); Sykehuset Innlandet HF (Other); Ullevaal University Hospital (Other); Sykehuset i Vestfold HF (Other); Sykehuset Ostfold (Other); Alesund Hospital (Other)
Responsible Party: Principal Investigator, Bjørn Naume, Principal investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBCG9; S-03032; S-03-01434
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: Disseminating tumor cells,breast cancer,docetaxel,adjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel (Experimental): Patients with presence of disseminated tumor cells in bone marrow after (no-taxane) epirubicin-containing adjuvant treatment receive 6 cycles of docetaxel (100 mg/m2) 3 qw.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 100 mg/m2 3 qw x 6
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to identify patients with persisting tumor cells after standard epirubicin-containing treatment to test a non-cross resistant chemotherapy regimen (docetaxel) for these patients, and to explore the analysis of disseminated tumor cells in bone marrow as a surrogate marker for clinical outcome.

DETAILED DESCRIPTION:
The presence of disseminating (or isolated) tumor cells (DTC/ITC) in bone marrow (BM) after completion of adjuvant chemotherapy for breast cancer is associated with poor prognosis. Methods for detection of DTC have potential as a tool for monitoring occult residual disease during follow up. Also, there exists potent chemotherapy proven to be effective when anthracycline-based chemotherapy fails (f.ex. docetaxel). Consequently, a study has been started to test DTC detection as a surrogate marker for clinical outcome in localized breast cancer patients, selected by the presence of DTC in BM after standard adjuvant chemotherapy, receiving secondary treatment with docetaxel. In brief, patients having received anthracycline-containing chemotherapy for localized breast cancer are candidates. After informed consent and no radiologic signs of distant metastasis, the first BM aspiration is performed at the end of radiotherapy or 8-12 weeks after the last chemotherapy cycle. The next BM aspiration is performed 6 months later. At that time point the BMs are analyzed for the presence of DTC. If DTC are present in the 6 months BM test (the first BM sample is for exploratory research purposes), 6 cycles of docetaxel are administered (3qw), followed by a third and forth BM analysis 1 month and 13 months after the end of chemotherapy. The patients receiving docetaxel with eradication of the DTC will be clinically compared to those with persistence of DTC after docetaxel treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer with node positive disease or high risk node negative disease (pT1c/T2GII-IIIN0, pT3N0, cT3N0). Patients < 35 years with pT1a-bN0G2-3.
2. Primary surgery for breast cancer completed
3. Completed 6 cycles of adjuvant (or neoadjuvant) chemotherapy containing anthracycline
4. Age ≥ 18 and < 70 years
5. Eastern Cooperative Oncology Group or WHO performance status < 2
6. Written informed consent prior to beginning protocol specific procedures
7. Laboratory requirements (within 5 weeks prior to end of radiation treatment or within 5 weeks prior to completion of baseline examinations):

   Neutrophils ≥ 1.1 10^9/l, Platelets ≥ 100 10^9/l, Hemoglobin ≥ 10 g/dl, ASAT and ALAT ≤ x 2.5 UNL (If ALP > 2.5 ≤ x 5 UNL, then ASAT and ALAT ≤ x 1.5 UNL), ALP ≤ x 5 UNL (If ASAT and ALAT > 1.5 ≤ x 2.5 UNL, then ALP ≤ 2.5 x UNL), Creatinine ≤ 175 umol/l
8. Completed staging analysis including chest X-ray, bone scintigraphy or MRI, liver ultrasound or liver CT scan

Exclusion Criteria:

1. Other (than breast carcinoma) earlier or concomitant carcinoma, except for skin and in situ cervix cancer
2. M1 breast cancer or locoregional recurrence of previously diagnosed breast cancer.
3. Earlier treatment with paclitaxel or docetaxel.
4. Pre-existing motor or sensory neurotoxicity of a severity ≥ grade 2 by NCI criteria (see appendix II)
5. Cardiac disease with symptoms classified as NYHA ≥ 2
6. Definite contraindications for the use of corticosteroids
7. Concurrent treatment with other experimental drugs
8. Concurrent treatment with any other anti-cancer therapy (except for endocrine therapy and trastuzumab)
9. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1128 (Actual)
Dates: Start 2003-10 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Disease free survival related to presence or absence of disseminated tumor cells | At approximately 8 years maximum FU

SECONDARY OUTCOMES:
Predictive value of primary tumor markers on effects of docetaxel | At approximately 8 years maximum FU
Explore markers on tumor cells in bone marrow that can predict the effect of docetaxel | At approximately of 8 years maximum FU

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Naume, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- RRHF, Oslo, Norway

REFERENCES:
- [Derived] Naume B, Synnestvedt M, Falk RS, Wiedswang G, Weyde K, Risberg T, Kersten C, Mjaaland I, Vindi L, Sommer HH, Saetersdal AB, Rypdal MC, Bendigtsen Schirmer C, Wist EA, Borgen E. Clinical outcome with correlation to disseminated tumor cell (DTC) status after DTC-guided secondary adjuvant treatment with docetaxel in early breast cancer. J Clin Oncol. 2014 Dec 1;32(34):3848-57. doi: 10.1200/JCO.2014.56.9327. Epub 2014 Nov 3. PMID 25366688
- [Derived] Gilje B, Nordgard O, Tjensvoll K, Borgen E, Synnestvedt M, Smaaland R, Naume B. Comparison of molecular and immunocytochemical methods for detection of disseminated tumor cells in bone marrow from early breast cancer patients. BMC Cancer. 2014 Jul 15;14:514. doi: 10.1186/1471-2407-14-514. PMID 25023626
- [Derived] Synnestvedt M, Borgen E, Wist E, Wiedswang G, Weyde K, Risberg T, Kersten C, Mjaaland I, Vindi L, Schirmer C, Nesland JM, Naume B. Disseminated tumor cells as selection marker and monitoring tool for secondary adjuvant treatment in early breast cancer. Descriptive results from an intervention study. BMC Cancer. 2012 Dec 22;12:616. doi: 10.1186/1471-2407-12-616. PMID 23259667